CLINICAL TRIAL: NCT01293708
Title: Realities, Expectations and Attitudes to Life Support Technologies in Intensive Care for Octogenarians:
Acronym: Realistic 80
Status: Completed | Type: Observational
Sponsor: Daren K. Heyland (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Daren K. Heyland, Dr. Daren Heyland, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Other Study IDs: R80
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Critically Ill
Keywords: Octogenarians; HRQOL; mortality; prospective observational; Elderly
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hospital Cohort: All 80+ year old that had had an ICU stay of >=24 hrs. Followed until hospital d/c
- Longitudinal Cohort: All 80+ year old that had had an ICU stay of >=24 hrs. Followed for 12 months

SUMMARY:
The purpose of this study is to understand the realities, expectations and attitudes of patients 80+ and their families about the use of life-sustaining technology, and to document the patient outcomes and family experiences associated with surviving and not surviving critical illness. Specifically in this project the investigators will determine the real outcomes of critical illness experienced by octogenarians.

DETAILED DESCRIPTION:
Seriously ill hospitalized elderly patients rate 'not being kept alive on prolonged life supports' as the most important aspect of good quality care at the end of life (EOL). Across Canada, large numbers of elderly patients near the EOL and their families are faced with decisions about whether or not to use mechanical ventilation or other forms of life support technology used in intensive care units (ICUs). The investigators do not know whether these patients and their families are informed about the realities of intensive care - that is, if they are aware of the likelihood of surviving a critical illness and the resultant health states. The outcomes of critical illness for this patient population and their families are unknown, despite the crucial importance of this information to guide clinical decision making. The goals of our research program are to understand the realities of critical care, and the expectations and attitudes of patients 80 years of age or older (80+) and their families about the use of life sustaining technology. Specifically, in this project, the investigators want to determine the realities or outcomes of surviving critical illness.

Our primary research question is:

1. What are the 12-month health-related quality of life (HRQOL), functional status, and survival of patients admitted to ICU who are 80+ years old?

   Our secondary research questions are:
2. Which patient characteristics are associated with 12-month HRQOL, functional status, and survival?
3. What is the satisfaction of family members with critical care, as measured by the Family Satisfaction in ICU (FS-ICU 24) instrument?
4. For patients surviving their ICU stay, what is the experience of family members caring for the patient during follow up, as measured by the Caregiver Reaction Assessment (CRA) instrument?
5. For patients who do not survive their ICU stay, what is the family satisfaction with EOL care, as measured using the CANHELP Satisfaction (Bereavement) instrument?
6. What is the health-related financial burden experienced by patients and their caregivers during their initial ICU hospitalization and up to 12 months after the index ICU admission?
7. What is the quality of decision making regarding the goals of care for an 80+ ICU patient?
8. What are the values that influence decisions about the goals of care for this population?

To answer these questions, the investigators are conducting a national, multicentre, cohort study of 800 patients age 80+ years who are admitted to Canadian ICUs. The investigators will follow these patients prospectively for 12 months to measure study outcomes. In addition, using novel instruments that the investigators have already developed and validated, the investigators will follow family members of these patients to document their experience as caregivers, their satisfaction with care of their relatives, and the financial implications of having a critically ill loved one. This quantitative project will be complemented by a separate qualitative study in the community setting to further understand the expectations and attitudes of persons over 80 years of age regarding the use of life sustaining technology. Data emerging from this work will inform important clinical decisions regarding critical care and EOL care for this aged population.

The investigators presume that the short- and long-term mortality of 80+ year olds admitted to Canadian ICUs will be high and that the self-reported health-related quality of life and functional status of survivors after hospital discharge will be low. The investigators anticipate that pre-morbid illnesses and functional status before admission to ICU will correlate with long-term clinical outcomes. The investigators are uncertain as to the psychological and financial burden experienced by families when a loved one is in the ICU and during the recovery phase; our study will be the first to furnish such important information. By using administrative databases to complement information already being collected in this study, the investigators will obtain a better understanding of the healthcare resource utilization and longer term survival of this cohort, and will be better positioned to offer effective ICU and follow-up care for this at-risk patient population.

ELIGIBILITY:
Inclusion Criteria:

* minimum stay in the ICU of 24 hrs
* patient is >=80 years old
* patient is a resident of Canada and has a permanent address in this country
* patient has an eligible family caregiver who has visited the patient at least once within 96 hours of the current ICU admission

Exclusion Criteria:

* family caregiver is <= 18
* family caregiver is paid to do so
* family caregivers that do not speak English or French
* previously enrolled

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 80+ year old admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 1504 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life (HRQOL) | 12 months
  To determine the 12 month HRQOL of 80+ year olds admitted to the ICU in Canada.

SECONDARY OUTCOMES:
To determine which patient characteristics are associated with 12-month HRQOL | 12 month
To determine which patient characteristics are associated with functional status. | 12 months
To determine which patient characteristics are associated with survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daren Heyland, MD, Study Chair — Clinical Evaluation Research Unit,, Kingston General Hospital
Locations (24):
- Canada (24):
  - Peter Lougheed Hospital, Calgary, Alberta
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - St.Paul's Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Vancouver, British Columbia
  - Victoria General Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Winnipeg Health Sciences Center, Winnipeg, Manitoba
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences, Toronto, Ontario
  - St. Michaels Hospital, Toronto, Ontario
  - Mount Sinai, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Hospital Maisonneuve-Rosemont, Montreal, Quebec
  - Hospital de Sacre-Coeur, Montreal, Quebec
  - Departement d'Anesthesie, Québec, Quebec
  - Hospital Laval, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Chin-Yee N, D'Egidio G, Thavorn K, Heyland D, Kyeremanteng K. Cost analysis of the very elderly admitted to intensive care units. Crit Care. 2017 May 16;21(1):109. doi: 10.1186/s13054-017-1689-y. PMID 28506243
- [Derived] Heyland DK, Garland A, Bagshaw SM, Cook D, Rockwood K, Stelfox HT, Dodek P, Fowler RA, Turgeon AF, Burns K, Muscedere J, Kutsogiannis J, Albert M, Mehta S, Jiang X, Day AG. Recovery after critical illness in patients aged 80 years or older: a multi-center prospective observational cohort study. Intensive Care Med. 2015 Nov;41(11):1911-20. doi: 10.1007/s00134-015-4028-2. Epub 2015 Aug 26. PMID 26306719
- [Derived] Heyland D, Cook D, Bagshaw SM, Garland A, Stelfox HT, Mehta S, Dodek P, Kutsogiannis J, Burns K, Muscedere J, Turgeon AF, Fowler R, Jiang X, Day AG; Canadian Critical Care Trials Group; Canadian Researchers at the End of Life Network. The Very Elderly Admitted to ICU: A Quality Finish? Crit Care Med. 2015 Jul;43(7):1352-60. doi: 10.1097/CCM.0000000000001024. PMID 25901550
- [Derived] Heyland DK, Dodek P, Mehta S, Cook D, Garland A, Stelfox HT, Bagshaw SM, Kutsogiannis DJ, Burns K, Muscedere J, Turgeon AF, Fowler R, Jiang X, Day AG; Canadian Critical Care Trials Group and Canadian Researchers at End of Life Network (CARENET). Admission of the very elderly to the intensive care unit: family members' perspectives on clinical decision-making from a multicenter cohort study. Palliat Med. 2015 Apr;29(4):324-35. doi: 10.1177/0269216314566060. Epub 2015 Feb 2. PMID 25645668